CLINICAL TRIAL: NCT06220643
Title: Prognosis and Effects of Ultrasound Guide Corticosteroid Injection with Progressive Resistance Exercise for Subacromial Bursitis: a Randomized Clinical Trial
Brief Title: Steroid Injection with Exercise for Subacromial Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, ShihWei Huang, Attending Physician, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202306022
Record Dates: First submitted 2023-12-14; First posted 2024-01-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Bursitis
MeSH Terms: interventions — Resistance Training; Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Echoguide steroid injection without exercise (only education) (Active Comparator): received 40mg triamcinolone acetonide 1cc plus 2cc lidocaine (1%) injected into the inflamed subacromial bursa with ultrasound guidance
  Interventions: Drug: triamcinolone acetonide plus lidocaine
- Echoguide steroid injection with exercise (Experimental): experimental group received 40mg triamcinolone acetonide 1cc plus 2cc lidocaine (1%) injected into the inflamed subacromial bursa with ultrasound guidance, and a 12-week elastic band progressive resistance exercise
  Interventions: Other: resistance exercise; Drug: triamcinolone acetonide plus lidocaine

INTERVENTIONS:
Other: resistance exercise — Progressive resistance exercise for 12 weeks
  Arms: Echoguide steroid injection with exercise
Drug: triamcinolone acetonide plus lidocaine — 40mg triamcinolone acetonide 1cc plus 2cc lidocaine (1%)
  Other Names: exercise education

SUMMARY:
Shoulder issues in middle-aged and elderly folks often stem from muscle and tendon degeneration, causing pain and limited movement. Current treatments like corticosteroid injections provide short-term relief for synovial bursitis, prompting repetitive injections. Combining these injections with resistance exercises, especially elastic bands, might extend relief. A study aims to test this by giving injections and a 12-week elastic band exercise program to one group, compared to injections alone in another. Assessments at 4, and 12 weeks post-injection will measure pain, motion, and functionality. Successful results could redefine treatment, reducing repetitive injections and enhancing life quality for those with shoulder problems.

DETAILED DESCRIPTION:
Shoulder activities are common among middle-aged and elderly individuals, often leading to degeneration of shoulder muscles and tendons. This degeneration causes instability, resulting in shoulder impingement syndrome and subsequent inflammation of the synovial bursa. Acute synovial bursitis leads to severe shoulder pain, limited movement, affecting daily life and work. Initial treatments like physical therapy and oral medication often fall short, necessitating corticosteroid injections into the subacromial bursa guided by ultrasound for effective relief. However, these injections often provide only short-term relief, leading to a need for repeated injections, causing concerns about side effects.

Previous research indicates that resistance-based exercises improve muscle strength and reduce shoulder tissue damage. Among these exercises, elastic band workouts are deemed safest for the elderly. Despite advancements in ultrasound-guided injections for subacromial bursitis, there's a scarcity of studies combining corticosteroid injections with progressive shoulder resistance exercises to prolong therapeutic effects.

This study aims to explore if progressive resistance exercises enhance and sustain the clinical benefits of ultrasound-guided corticosteroid injections in subacromial bursitis. It's a randomized double-single-blind study wherein the experimental group receives ultrasound-guided injections of 40mg triamcinolone acetonide and 2cc lidocaine into the inflamed bursa and undergoes a 12-week course of elastic band progressive resistance exercises. The control group only receives ultrasound-guided injections. Evaluators remain unaware of the group assignments. Parameters like VAS , ROM, and SPADI are assessed at 4, and 12 weeks post-injection.

This research seeks to ascertain whether combining corticosteroid injections with progressive resistance exercises prolongs the efficacy of treatment for subacromial bursitis. If successful, it could offer a novel approach to managing this condition, potentially reducing the need for repeated injections and improving the overall quality of life for middle-aged and elderly individuals affected by shoulder issues.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of subacromial bursitis of shoulder

Exclusion Criteria:

* history of shoulder shoulder and operation history
* comorbid with adhesive capsulitis or rotator cuff tear
* received local injection of shoulder with steroid, hypertonic dextrose, hyaluronic acid or platelet-rich plasma in recent 6 months

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Day 0, Month 1, Month 3
  The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with ADLs requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items.
Visual Analogue Scale (VAS) | Day 0, Month 1, Month 3
  pain score from 0~10, 0 means no pain, and 10 means extreme pain

SECONDARY OUTCOMES:
pain free range of motion | Day 0, Month 1, Month 3
  Shoulder range of motion of flexion, extension, abduction, internal rotation, external rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City, Zhonghe Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No